CLINICAL TRIAL: NCT05157581
Title: Open Label, Single-cohort, and Multi-center Phase II Study Evaluating Tumor-specific Immunity After Extracorporeal Photopheresis in Patients With Sézary Syndrome at Single-cell Resolution
Brief Title: Extracorporeal Photopheresis in Sezary Syndrome
Acronym: ECP
Status: Recruiting | Type: Observational
Sponsor: Oleg E. Akilov, MD, PhD (Other)
Collaborators: Therakos (Industry)
Responsible Party: Sponsor-Investigator, Oleg E. Akilov, MD, PhD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY21100115
Record Dates: First submitted 2021-11-16; First posted 2021-12-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sezary Syndrome
Keywords: extracorporeal photopheresis
MeSH Terms: conditions — Sezary Syndrome | interventions — Photopheresis; Methoxsalen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Sezary Syndrome: 20 subjects with Sezary Syndrome will comprise the single arm of this study
  Interventions: Device: Extracorporeal photopheresis (ECP); Drug: Methoxsalen Injection

INTERVENTIONS:
Device: Extracorporeal photopheresis (ECP) — Extracorporeal photopheresis is a process that exposes a collection of white blood cells and plasma to a light sensitizing agent, methoxsalen, and returns that compartment to the body.
  Other Names: ECP; photopheresis
Drug: Methoxsalen Injection — Methoxsalen is a light-sensitizing sterile compound added to the collected white blood cells and plasma during ECP.
  Other Names: Uvadex

SUMMARY:
The primary endpoint is to determine if ECP induces a decrease in % of tumor cells after treatment. 20 patients with Sezary Syndrome will receive ECP weekly x4, then bi-weekly for 5 months. Each patient will donate 5 samples to determine immune responses in peripheral blood. Additional clinical assessments will be a modified skin weighted assessment and flow cytometry at baseline and months 3 and 6. A CT scan will be obtained at baseline and only repeated if pathology is present at baseline. The tumor microenvironment will be studied by comparing transcriptomics of the blood samples before, 1 day after first ECP treatment, cycle 1, 1, 3 and 6 months after ECP treatment by scRNAseq (5 samples total per patient ).

DETAILED DESCRIPTION:
Cutaneous T-cell lymphoma (CTCL) is a group of skin lymphomas in which malignant lymphocytes infiltrate the skin and, in the later stages, spread to the lymph nodes and blood (leukemia). In the early stages, CTCL generally has a slow course, but in advanced diseases, such as Sezary syndrome (the leukemic form of the disease), there is rapid deterioration. Sezary syndrome is an end-stage variant of CTCL with a mean survival of 1.5 years despite aggressive therapies. Treatment options for the advanced disease are severely limited.

In this study, informed consent will be offered to patients who are candidates for standard of care ECP and have a diagnosis of Sezary Syndrome. Participating patients will undergo ECP twice weekly for 4 weeks then twice monthly for 5 more months (month 6 of therapy). Research blood samples to assess immune responses will be obtained from a blood draw at baseline (before starting ECP), one day after first ECP, and at months 1, 3, and 6. Standard of care assessments to determine the objective response will include measurement of skin tumor burden (mSWAT), blood tumor burden (flow cytometry) and CT scan at baseline and only repeated at month 3 and 6 if lymph node or visceral (organ) involvement identified at baseline.

The investigators propose to establish changes in the tumor microenvironment after ECP, compare transcriptomic differences in malignant lymphocytes, monocytes, DC, and CD8 effectors before and after ECP to test the hypothesis that anti-tumor immune responses can be induced by ECP. We will employ a highly innovative technology such as single-cell RNA sequencing (scRNAseq) coupled with TCR sequencing to characterize ECP-related change in malignant cells utilizing a custom gene set and validate the single-cell protein data by antibody-oligo conjugates. To better understand the relevance of biomarker changes to disease progression, the observed ECP-related changes in tumor microenvironment will be correlated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an established diagnosis of Sezary syndrome (stage IVA1)
2. Patients amenable for ECP
3. The patient must have a minimum wash-out period of 3 weeks between the last dose of prior systemic therapy
4. Patients should have recovered from all adverse events related to prior therapy to ≤ grade 1
5. Signed informed consent form prior to any protocol-specific procedures.

Exclusion Criteria:

1. Visceral metastasis of lymphoma
2. Concomitant administration of radiotherapy or systemic anti-cancer therapy including but not restricted to: chemotherapy, biological agents, or immunotherapy
3. Patients with known NCI CTCAE grade 3 or higher active systemic or cutaneous viral, bacterial, or fungal infection.
4. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment and/or comply with study protocol.
5. Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent document.
6. Patients with known allergy to Methoxsalen or heparin (as part of SOC ECP procedure).
7. Patients who are pregnant. -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Sezary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in tumor-specific immunity | Up to 3 months post baseline
  Evaluate immune responses post ECP using innovative technology such as single-cell RNA sequencing (scRNAseq) coupled with TCR sequencing to characterize ECP-related change in malignant cells
Change from baseline in tumor-specific immunity | Up to 6 months post baseline
  Evaluate immune responses post ECP using innovative technology such as single-cell RNA sequencing (scRNAseq) coupled with TCR sequencing to characterize ECP-related change in malignant cells

SECONDARY OUTCOMES:
Change from baseline in the objective response rate for ECP therapy | Up to 3 months post baseline
  .Evaluate response in skin and blood using a modified skin weighted assessment tool that assess the tumor burden in the skin and blood flow cytometry that assesses the tumor burden in the blood. If tumor burden detected internally (visceral) or in the lymph nodes at baseline, follow up CT scans will be used to evaluate lymph nodal and/or visceral response. Response rate is defined as 50% or greater decrease in skin, lymph node/visceral, or blood tumor burden
Change from baseline in the objective response rate for ECP therapy | Up to 6 months post baseline
  .Evaluate response in skin and blood using a modified skin weighted assessment tool that assess the tumor burden in the skin and blood flow cytometry that assesses the tumor burden in the blood. If tumor burden detected internally (visceral) or in the lymph nodes at baseline, follow up CT scans will be used to evaluate lymph nodal and/or visceral response. Response rate is defined as 50% or greater decrease in skin, lymph node/visceral, or blood tumor burden

OTHER OUTCOMES:
Change from baseline in the objective response rate by disease compartment | Up to 3 months post baseline
  Evaluation of objective responses separated out by each subgroup of potential involvement (blood, skin, lymph nodes,and viscera (if present).
Change from baseline in the objective response rate by disease compartment | Up to 6 months post baseline
  Evaluation of objective responses separated out by each subgroup of potential involvement (blood, skin, lymph nodes,and viscera (if present).
Correlation of clinical responses and changes in tumor microenvironment in the blood. | Up to 6 months post baseline
  Technology using scRNAseq to analyze the blood microenvironment will be correlated with the clinical responses observed.

CONTACTS AND LOCATIONS:
Overall Officials: Oleg E Akilov, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Cutaneous Translational Research Program - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ying Z, Shiue L, Park K, Kollet J, Bijani P, Goswami M, Duvic M, Ni X. Blood transcriptional profiling reveals IL-1 and integrin signaling pathways associated with clinical response to extracorporeal photopheresis in patients with leukemic cutaneous T-cell lymphoma. Oncotarget. 2019 May 7;10(34):3183-3197. doi: 10.18632/oncotarget.26900. eCollection 2019 May 7. PMID 31139332
- [Background] Zic JA. Extracorporeal Photopheresis in the Treatment of Mycosis Fungoides and Sezary Syndrome. Dermatol Clin. 2015 Oct;33(4):765-76. doi: 10.1016/j.det.2015.05.011. Epub 2015 Jul 29. PMID 26433848
- [Background] Spary LK, Al-Taei S, Salimu J, Cook AD, Ager A, Watson HA, Clayton A, Staffurth J, Mason MD, Tabi Z. Enhancement of T cell responses as a result of synergy between lower doses of radiation and T cell stimulation. J Immunol. 2014 Apr 1;192(7):3101-10. doi: 10.4049/jimmunol.1302736. Epub 2014 Mar 5. PMID 24600032
- [Background] Curion F, Handel AE, Attar M, Gallone G, Bowden R, Cader MZ, Clark MB. Targeted RNA sequencing enhances gene expression profiling of ultra-low input samples. RNA Biol. 2020 Dec;17(12):1741-1753. doi: 10.1080/15476286.2020.1777768. Epub 2020 Jun 28. PMID 32597303